CLINICAL TRIAL: NCT01243879
Title: The Effect of Food Stimuli on the Calorie Restriction Response in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Center for Medical Systems Biology (Unknown); Roba Metals BV, IJsselstein (Unknown)
Responsible Party: Principal Investigator, Hanno Pijl, Prof. dr. H. Pijl, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P08.077
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Calorie Restriction; Aging
Keywords: fasting; starvation; calorie restriction; fMRI
MeSH Terms: conditions — Fasting; Starvation | interventions — Vision, Ocular; Stimuli Responsive Polymers

ARMS (2):
- Fasting with stimuli (Active Comparator): Fasting in the presence of food-related stimuli
  Interventions: Other: Stimuli of food smell and vision
- Fasting without stimuli (Sham Comparator): Fasting in the absence of food-related stimuli
  Interventions: Other: No stimuli of food smell and vision

INTERVENTIONS:
Other: Stimuli of food smell and vision — 60 hours of starvation (fasting) in the presence or absence of visual and odorous food cues
  Other Names: Stimuli
  Arms: Fasting with stimuli
Other: No stimuli of food smell and vision — 60 hours of starvation (fasting) in the presence or absence of visual and odorous food cues
  Other Names: No Stimuli
  Arms: Fasting without stimuli

SUMMARY:
Calorie restriction extends life span and prevents aging-related diseases in several species. Odorants from live yeast restrain the beneficial effects of calorie restriction in Drosophila Melanogaster. The investigators hypothesize that visual and odorous food stimuli impact the neuroendocrine and metabolic response to starvation in healthy humans.

In this randomized cross-over intervention study 12 healthy, young men will fast twice for 60-hours in the presence or absence of food-related visual and odorous stimuli. At baseline and on the last morning of each intervention an oral glucose tolerance test (OGTT) will be performed. During the OGTT blood is sampled and hypothalamic neuronal activity is measured by functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male volunteers
* Age > 18 years and < 70 years
* Body mass index (BMI) > 20 kg/m2 and < 25 kg/m2
* Fasting serum glucose (FSG) < 6.1 mmol/L

Exclusion Criteria:

* Any significant chronic of hereditary disease (including renal, hepatic or endocrine disease)
* Any significant abnormal laboratory results found during the medical screening procedure
* Any use of medication (except for NSAID)
* Anosmia or any other (acquired) loss of olfaction (ea. rhinitis)
* Recent weight changes or attempts to loose weight (> 3 kg weight gain or loss, within the last 3 months)
* Difficulties to insert an intravenous catheter
* Smoking
* MRI contraindications
* Recent blood donation (within the last 3 months)
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Endocrine and metabolic outcomes | 4 weeks
  The effects of odors and / or visual stimuli of food in subjects after 60h of starvation on: endocrine parameters, metabolic parameters, anthropometric parameters

SECONDARY OUTCOMES:
functional Magnetic Resonance Imaging | 4 weeks
  The effects of odors and / or visual stimuli of food in subjects after 60h of starvation on hypothalamic neuronal activity